CLINICAL TRIAL: NCT04755153
Title: Community Intervention to Reduce CardiovascuLar Disease in Chicago
Acronym: CIRCL-Chicago
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Utah (Other); Pastors 4 PCOR (Unknown)
Responsible Party: Principal Investigator, Justin D. Smith, Adjunct Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00212622
Record Dates: First submitted 2021-02-03; First posted 2021-02-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Practice Facilitation (Experimental): Practice Facilitation to support implementation of the Kaiser Blood Pressure Control Bundle
  Interventions: Other: Practice Facilitation
- Non-Practice Facilitation (Active Comparator): implementation of the Kaiser Blood Pressure Control Bundle without Practice Facilitation
  Interventions: Other: Non-Practice Facilitation

INTERVENTIONS:
Other: Practice Facilitation — Tailored interventions provided by a trained Practice Facilitator
  Arms: Practice Facilitation
Other: Non-Practice Facilitation — Implementation support without using Practice Facilitation
  Arms: Non-Practice Facilitation

SUMMARY:
Hypertension affects 1 in every 3 adults in the US and contributes to 410,000 deaths annually. Hypertension and its associated complications disproportionately affect minority populations living in urban areas. In Chicago, health status indicators show worsening disparities between black and white residents, with the highest rates of hypertension, heart disease, and stroke clustering in the predominantly black South and West Sides. Kaiser Permanente demonstrated that a bundle of evidence-based interventions implemented within a large, integrated health system in Northern California significantly increased blood pressure control rates. However, it is unclear whether a health system centered intervention can be adapted to other settings, particularly under-resourced urban communities. Therefore, the overall goal is to support a community-centered design and adaptation of the Kaiser bundle. The investigative team will adapt the delivery model of the Kaiser bundle to be centered within churches within the South Side of Chicago, one of the most medically underserved communities in the United States. The proposed interventions are the same as in the Kaiser bundle (e.g., registry/audit and feedback, simplified treatment regimens, accurate Blood Pressure measurement) but implementation of the components of the bundle will be adapted for delivery in the community. The intervention will be carried out by local community health workers and ministry facilitators, with health clinics and hospitals in the community as support, all connected through a common data platform.

Thus, the proposed project will identify the best strategies to support adoption, implementation with fidelity, and sustainability of the Kaiser bundle in the community setting. The proposed study will follow the Exploration, Preparation, Implementation and Sustainment (EPIS) process model and implementation is rigorously evaluated using a multimethod approach to the Reach, Effectiveness, Adoption, Implementation, and Maintenance (REAIM) evaluation framework. The specific aims are: Aim 1: Convene community stakeholders in order to adapt implementation strategies using the Dynamic Adaptation Process model. Aim 2: Design, implement, and evaluate pilot projects in order to optimize implementation strategies within the target community. Aim 3: Implement, test and evaluate an adapted implementation strategy to control hypertension through faith-based organizations in the South Side of Chicago. The study uses a hybrid Type 3 effectiveness-implementation design based within one primary community area (South Side Chicago) and in two settings (church and clinic). The overall study outcomes reach (implementation) and blood pressure (clinical effectiveness). Aim 4: Disseminate findings internally to community stakeholders and externally through creation of community implementation toolkits.

ELIGIBILITY:
Inclusion Criteria:

* Community: patients w/in participating clinics (by clinic location in community) OR within participating churches (by location in community)
* Age: adults (18-89 y/o)

Exclusion Criteria:

* Children less that 18 years of age

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 3-6 months per patient
  The investigators will examine change in systolic blood pressure measured via automatic and manual devices as a result of participating in the intervention

SECONDARY OUTCOMES:
Feasibility of implementation | 2 years
  The investigators will evaluate stakeholder perceptions of the feasibility of the Kaiser BP Bundle and how it is being implemented after an iterative community-based adaptation process prior to and during the trial. This measure will use the validated Feasibility of Implementation (FIM) scale (Weiner et al. 2017) which contains 3-items rated on a scale of 1-5 (range: 3-15) with higher scores indicating greater feasibility.
Acceptability of Intervention Measure | 2 years
  The investigators will evaluate stakeholder perceptions of the acceptability of delivering the Kaiser BP Bundle after an iterative community-based adaptation process prior to and during the trial. This measure will use the validated Acceptability of Intervention Measure (AIM) (Weiner et al. 2017) which contains 3-items rated on a scale of 1-5 (range: 3-15) with higher scores indicating greater acceptability.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Pastors4PCOR, Chicago, Illinois
  - Access Community Health Network, Chicago, Illinois
  - Advocate Aurora Health, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Available by request 1 year after completion of enrollment
Time Frame: Available by request 1 year after completion of enrollment

REFERENCES:
- [Derived] Smith JD, Carroll AJ, Tedla YG, Sanuade OA, Merle JL, Heinrich J, Bannon J, Abramsohn EM, Ahmad FS, Lazar D, Lindau ST, McHugh MC, Khatib R, Donovan R, Pinkerton EA, Rosul LL, Walunas TL, Watson R, Ganbote T, Kandula N, Youmans QR, Davis P, Kho AN. Community intervention to reduce cardiovascular disease in Chicago (CIRCL-Chicago): protocol for a type 3 hybrid effectiveness-implementation study using a parallel cluster-randomized trial design. Implement Sci. 2025 May 5;20(1):19. doi: 10.1186/s13012-025-01431-w. PMID 40325453

DOCUMENTS (1):
  • Informed Consent Form (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT04755153/ICF_000.pdf